CLINICAL TRIAL: NCT01760278
Title: Assessment of Implantation Potential of Embryos Cultured by Time-lapse Technology (Embryoscope) Before Transfer in In-vitro Fertilization (IVF) / Intracytoplasmic Sperm Injection (ICSI) Cycles: A Randomized Control Study.
Brief Title: Assessment of Implantation Potential of Embryos by Time-lapse Technology
Acronym: Embryoscope
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bloom IVF and Fertility Centre (Other)
Collaborators: Padmashree Dr. D. Y. Patil Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Time-lapse monitoring; Study of embryo morphokinetics (Other: Bloom IVFand Fertility Centre)
Record Dates: First submitted 2012-12-26; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Embryo/Fetus Death; Blastocyst Disintegration; Aneuploidy; Complication of Implant; Chemical Pregnancy
Keywords: Time-lapse monitoring of embryos.; Embryoscope; IVF-ET/ICSI; Cetrorelix; Gonal-F
MeSH Terms: conditions — Stillbirth; Embryo Loss; Aneuploidy | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Arm (Experimental): Subjects would receive recombinant Follicle Stimulating Hormone (rFSH) by S.C. injection 150 - 225 IU/day for 9 days. The embryos of subjects would be cultured by time-lapse imagery technique (embryoscope) and analysis would be done using patients receive rFSH (Gonembryo viewer equipped with latest software.
  Interventions: Drug: recombinant Follicle Stimulating Hormone (rFSH)
- Control Arm (Active Comparator): Subjects would receive recombinant Follicle Stimulating Hormone (rFSH) by S.C. injection 150 - 225 IU/day for 9 days. The embryos of subjects would be cultured in conventional culture environment and analysis would be done using established subjective morphological criteria.
  Interventions: Drug: recombinant Follicle Stimulating Hormone (rFSH)

INTERVENTIONS:
Drug: recombinant Follicle Stimulating Hormone (rFSH) — There are two arms of the study. The Study arm and the Control arm. In each arm, subjects, after randomization, will be stimulated with rFSH 225IU/day.
  On day 6, Cetrorelix 0.25mg/day to be added till the day of Ovitrell. Thereafter, ovum pick-up and embryo transfer to be done. Six weeks after transfer clinical pregnancy identified which will be the end-point of the study.
  Other Names: Gonal-F; Progesterone vaginal; Ovitrell 250mcg; Cetrorelix 0.25 mg

SUMMARY:
1. Culture conditions of developing embryos are highly controlled in the Embryoscope and are monitored by Time-lapse videography to produce 3D images at different stages.This cannot be done under conventional culture conditions.
2. The 3D images thus produced,are analysed with the help of Embryoviewer, a part of the Embryoscope,through latest software.
3. Embryoviewer also identifies embryos for transfer, freezing and to be discarded.

DETAILED DESCRIPTION:
1. There will be two arms of the study. The Study arm in which embryos of patients will be cultured in the Embryoscope. The control arm in which the embryos of patients will be cultured under conventional conditions.
2. Embryos to be transferred will be identified by the Embryoviewer in the Study arm and the ones in the control arm will be identified by established subjective morphological criteria.
3. Embryos with definite implantation potential will be transferred in both arms.
4. Embryos not transferred will be frozen and/or discarded in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. Women of age 21-39 yrs.
2. Basal FSH < 12mIU/ml
3. Anterior mullerian hormone(AMH) > 1.0 ng/ML
4. Antral follicle count (AFC) > 8
5. Body mass index (BMI) < 35 mt2/kg
6. Estradiol (E2) < 50PG/ML

Exclusion Criteria:

1. Women with one ovary.
2. Women in whom both ovaries are not seen on ultrasonography.
3. Women with too small uterine cavity.
4. Women with history of recurrent pregnancy loss
5. Women with systemic lupus erythematosus (SLE), Nephrotic syndrome, Meyer Rocky Tansky Kustner Hammer(MRKH) syndrome,etc.
6. Human immunodeficiency virus (HIV) I and II positive women.

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
No.of top quality embryos produced in both the arms, study arm and control arm. | 2 weeks
  1. 4-cell embryos on day 2 of fertilization in both,Study arm and Control arm.
  2. 8-cell embryos on day 3 of fertilization in both Study arm and Control arm.
  3. Blastocyst embryos on day 5 or day 6 of fertilization in both Study arm and Control arm.

SECONDARY OUTCOMES:
Clinical pregnancy | 6 weeks after embryo transfer (ET)
  Clinical pregnancy will be identified by presence of gestational sac(s) and fetal heart-beat by transvaginal ultrasonography in sixth week after embryo transfer.

OTHER OUTCOMES:
No. of mature M2 oocytes obtained | 2 weeks
  Mature oocyte identified by presence of polar body, fluffy granulosa cells surrounded by corona radiata.

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh D Pai, M.D., Principal Investigator — Bloom IVF and Fertility Centre; Manchi R Bharucha, Ph.D., Study Director — Bloom IVF and Fertility Centre
Locations (1):
- Lilavati Hospital and Research Center, IVF department, Mumbai, Maharashtra, India

REFERENCES:
- [Result] Lemmen JG, Agerholm I, Ziebe S. Kinetic markers of human embryo quality using time-lapse recordings of IVF/ICSI-fertilized oocytes. Reprod Biomed Online. 2008 Sep;17(3):385-91. doi: 10.1016/s1472-6483(10)60222-2. PMID 18765009